CLINICAL TRIAL: NCT00980252
Title: Medication Adherence in Schizophrenia: Development of a CBT-Based Intervention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Illinois at Chicago (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Peter Weiden, Professor, University of Illinois at Chicago
Allocation: Randomized | Model: Parallel | Masking: Triple
Other Study IDs: R34MH080978 (NIH); R34MH080978 (NIH); R34MH080978-01A2 (NIH); DSIR 83-AT
Record Dates: First submitted 2009-09-18; First posted 2009-09-21 (Estimated); Last update posted 2014-06-16 (Estimated); Status verified 2014-06

CONDITIONS: Schizophrenia; Psychotic Disorders
Keywords: Schizophrenia; Cognitive Behavioral Therapy; Compliance; Medication Adherence; Psychotic Disorders; Mental Disorders; Outcomes; Psychoeducation; Adherence Attitudes; Intervention; Nonadherence; Schizophrenia and Disorders with Psychotic Features
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders; Patient Compliance; Medication Adherence; Mental Disorders; Schizophrenia Spectrum and Other Psychotic Disorders | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (1):
- CBT (Experimental): UK-based intervention
  Interventions: Behavioral: Cognitive Behavioral Therapy

INTERVENTIONS:
Behavioral: Cognitive Behavioral Therapy — Brief intervention of Cognitive Behavioral Therapy sessions compared to Team Solutions

SUMMARY:
This is a randomized pilot study of an intervention based on principles of Cognitive Behavioral Therapy (CBT). This intervention is the Health Dialogue Intervention (HDI) and will be compared to a traditional medical model of psychoeducation known as Team Solutions (TS) for first-episode schizophrenia patients. Outcomes include the acceptance of HDI and TS, compare adherence attitudes at the end of the treatment intervention, and to compare the time until the first episode of nonadherence.

DETAILED DESCRIPTION:
Overview: Many people recovering from first-episode schizophrenia typically respond very well to their initial course of antipsychotic medications; however, studies indicate that nonadherence rates soar as high as 90% in the first year and do not improve over time. To date, there is no effective psychosocial intervention that improves adherence or reduces the adverse consequences of nonadherence after it occurs. Thus, it is imperative to develop a new intervention to improve medication adherence and improve clinical outcomes in patients recovering from first-episode schizophrenia.

This study is to pilot an intervention specifically suited for patients with first-episode schizophrenia based on the principles of Cognitive Behavioral Therapy (CBT). This is to focus on adherence from the perspective of the patient.

Methods: This study compares the effectiveness of a standard psychoeducation program [Team Solutions (TS)] to a CBT approach known as the Health Dialogue Intervention (HDI). Consenting patients will receive a 4 week stabilization assessment period and then be randomized to a prospective, random-assignment study comparing the effectiveness of TS to HDI to improve medication adherence of patients recovering from first-episode schizophrenia.

ELIGIBILITY:
There is a 2 step inclusion/exclusion criteria, the first being for assessing overall eligibility to enter the study, and then, for continued outpatient treatment for schizophrenia, schizophreniform disorder, or schizoaffective disorder.

Inclusion criteria for entry into the Evaluation Phase:

1. Between 16-45 years of age
2. A provisional clinical diagnosis of schizophreniform disorder, schizophrenia, or schizoaffective disorder in last 6 months
3. Discharge from inpatient unit for treatment of psychotic symptoms must have occurred in the last 6 months, or, if never hospitalized, initial treatment started in the last 6 months
4. Able to fully participate in the informed consent process
5. The patient is judged to be an appropriate candidate for ongoing outpatient follow-up at the First-episode Treatment Program at the Psychotic Disorders Program at UIC

Exclusion criteria for the Evaluation Phase:

1. Unable to understand informed consent process
2. A history of nonresponse to prior antipsychotic trials such that long-term inpatient treatment or clozapine will be recommended
3. Prior treatment with clozapine
4. Discharge from inpatient treatment for psychotic symptoms, initial treatment, or provisional diagnosis of schizophrenia, schizoaffective disorder, or schizophreniform occurred more than 6 months from enrollment into the evaluation phase
5. Pregnancy or stated goal to become pregnant
6. Will not be living close enough to the medical center to return for follow-up visits or assessments
7. History of geographic instability such that it is judged unlikely that patient will reside in the area
8. Currently under arrest for a felony, or an arrest is deemed likely in the near future
9. Currently receiving medication over objection by court order
10. Currently receiving treatment in another research protocol

Inclusion Criteria for the Treatment Intervention Phase:

1. Willingness to transition to receive evaluation and future pharmacologic treatment at the Psychotic Disorders Program at UIC
2. Has capacity to understand the risks and benefits of participating in a randomized psychosocial trial
3. Willingness to sign informed consent to go into the Treatment Intervention Phase
4. Is able to complete a post-test for understanding the nature of the study and what it entails, and the potential risks and benefits of study participation
5. Is willing to have therapy sessions recorded for fidelity assessments
6. Is willing to receive follow-up independent assessments of adherence status, including separate interviews with trained independent raters, and our contacting the outpatient pharmacy for pharmacy refill records

Exclusion criteria for Treatment Intervention Phase:

1. Diagnosis or inpatient treatment for psychotic symptoms occurred more than 6 months from date of enrollment into evaluation phase
2. Acutely psychotic individuals may not participate because therapy will not benefit if symptoms are too severe
3. Has dropped out of the treatment program and cannot be located for follow-up appointments
4. Stated refusal to come for to at least one clinical evaluation appointment at the PDP, or has been a "no show" for at least three consecutive appointments
5. Judged to be at significant and imminent risk of harm to self or others*
6. Ongoing active substance or alcohol use that is not controlled during the Evaluation Phase, along with refusal of referral to a "dual diagnosis" treatment program for substance abuse problems
7. Remains enrolled in another research protocol at UIC*
8. Unwilling to consider any additional psychotherapeutic intervention above and beyond coming in to the service for medication management appointment
9. Baseline PANSS total score ≥ 90, or has a individual PANSS item of conceptual disorganization (item P2), excitement (P4), or hostility (P7) that is ≥ 5 (moderately severe)*
10. Judged to require additional concrete case management services to support medication adherence*
11. Receives antipsychotics under coercive conditions (e.g. inpatient or outpatient commitment)*

Note: The exclusion criteria (*) may be present during some parts of the Evaluation Phase and would need to be resolved within the 4 week time period permitted for the Evaluation Phase prior to the Treatment Intervention Phase of study entry.

Ages: 16 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 34 (Actual)
Dates: Start 2009-11; Primary Completion 2012-12 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
1. Acceptance of therapeutic intervention as measured by number of sessions attended. 2. Difference in adherence behavior as measured by duration of antipsychotic treatment during follow up (ASV). 3. Differences in adherence attitudes (ROMI). | Completion of Study

SECONDARY OUTCOMES:
1. Compare the course of symptoms and relapse of patients in HDI to those in the TS. | Completion of Study

CONTACTS AND LOCATIONS:
Overall Officials: Peter J. Weiden, M.D., Principal Investigator — University of Illinois at Chicago
Locations (1):
- University of Illinois at Chicago, Chicago, Illinois, United States